CLINICAL TRIAL: NCT02273115
Title: Foley With Oxytocin Versus Foley no Oxytocin for Induction of Labor (NOFOX): a Randomized Control Trial
Brief Title: Foley With Oxytocin Versus Foley no Oxytocin for Induction of Labor
Acronym: NOFOX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Collaborators: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Corina Schoen, Maternal Fetal Medicine Fellow, Christiana Care Health Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCC-34107
Record Dates: First submitted 2014-10-20; First posted 2014-10-23 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Labor; Forced or Induced, Affecting Fetus or Newborn
Keywords: induction; Foley catheter; oxytocin
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nulliparous - Foley only (Active Comparator): Nulliparous women randomized to receive Foley only treatment will have a 20 French latex or silicone Foley catheter placed by the provider in the method they are most comfortable (direct visualization or indirectly). Balloons will have the ability to accommodate up to 80 ml of fluid to avoid rupture. The Foley balloon with be instilled with 60 ml of saline. The end of the catheter is then taped to the medial aspect of the patient's thigh on tension. No additional ripening agents or oxytocin will be administered while the Foley is in place. If spontaneous expulsion has not occurred, the Foley will be removed after 12 hours. Oxytocin will be administered per Christiana Care protocol after Foley removal.
  Interventions: Device: Transcervical Foley catheter
- Nulliparous - Foley and oxytocin (Active Comparator): Nulliparous women randomized to receive Foley and oxytocin treatment will have a 20 French latex or silicone Foley catheter placed by the provider in the method they are most comfortable (direct visualization or indirectly). Balloons will have the ability to accommodate up to 80 ml of fluid to avoid rupture. The Foley balloon with be instilled with 60 ml of saline. The end of the catheter is then taped to the medial aspect of the patient's thigh on tension. If spontaneous expulsion has not occurred, the Foley will be removed after 12 hours. Oxytocin will be administered per Christiana Care protocol immediately after Foley placement.
  Interventions: Drug: Oxytocin; Device: Transcervical Foley catheter
- Multi(primi)parous - Foley only (Active Comparator): Multiparous and primiparous women randomized to receive Foley only treatment will have a 20 French latex or silicone Foley catheter placed by the provider in the method they are most comfortable (direct visualization or indirectly). Balloons will have the ability to accommodate up to 80 ml of fluid to avoid rupture. The Foley balloon with be instilled with 60 ml of saline. The end of the catheter is then taped to the medial aspect of the patient's thigh on tension. No additional ripening agents or oxytocin will be administered while the Foley is in place. If spontaneous expulsion has not occurred, the Foley will be removed after 12 hours. Oxytocin will be administered per Christiana Care protocol after Foley removal.
  Interventions: Device: Transcervical Foley catheter
- Multi(primi)parous - Foley and oxytocin (Active Comparator): Multiparous and primiparous women randomized to receive Foley and oxytocin treatment will have a 20 French latex or silicone Foley catheter placed by the provider in the method they are most comfortable (direct visualization or indirectly). Balloons will have the ability to accommodate up to 80 ml of fluid to avoid rupture. The Foley balloon with be instilled with 60 ml of saline. The end of the catheter is then taped to the medial aspect of the patient's thigh on tension. If spontaneous expulsion has not occurred, the Foley will be removed after 12 hours. Oxytocin will be administered per Christiana Care protocol immediately after Foley placement.
  Interventions: Drug: Oxytocin; Device: Transcervical Foley catheter

INTERVENTIONS:
Drug: Oxytocin
  Arms: Multi(primi)parous - Foley and oxytocin; Nulliparous - Foley and oxytocin
Device: Transcervical Foley catheter
  Other Names: Transcervical Foley balloon

SUMMARY:
The overall purpose of this study is to determine if adding oxytocin to a Foley catheter for induction of labor will increase the rate of delivery within 24 hours stratified by parity.

DETAILED DESCRIPTION:
This is a multi-center, open-label, randomized study. Women with a singleton, vertex gestation between 24-42 weeks gestations presenting for labor induction will be offered participation in this study. Patients who receive prenatal care at Christiana Care may be approached if an induction of labor is scheduled and consented at their prenatal visit. All indications for induction will be included except those specifically mentioned as exclusion criteria. Any contraindication for vaginal delivery would exclude the subject. After informed consent is obtained, the Foley catheter will be placed and the subject will be randomized to receive oxytocin (study group) or not (control group). After Foley catheter removal or expulsion, the remainder of the induction course was left to the discretion of the primary provider. Prior to randomization, the subject will be placed into the nulliparous or multiparous group.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Pregnant, singleton gestation, vertex presentation
* Admitted for induction of labor between gestational ages 24 - 42 weeks
* Bishop score <6

Exclusion Criteria:

* Multiple gestation
* Non-vertex presentation
* Latex allergy or latex-free Foley catheter to be placed
* Fetal death
* Anomalous fetus
* Placenta/vasa previa
* Placental abruption (known or suspected)
* Intrapartum bleeding
* Non-reassuring fetal tracing with following criteria: category III tracing, OR minimal variability AND decelerations of any kind, OR late decelerations occurring >50% of contractions
* 2 or more previous cesarean section, myomectomy, or classical cesarean
* Need to use ripening agents prior to Foley placement
* Spontaneous labor
* Active genital herpes
* Inability to consent
* Any contraindication to a vaginal delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2014-10; Primary Completion 2016-09-11 (Actual); Study Completion 2016-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corina Schoen, MD, Principal Investigator — Sidney Kimmel Medical College at Thomas Jefferson University
Locations (2):
- United States (2):
  - Christiana Care Health Services, Newark, Delaware
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bujold E, Blackwell SC, Gauthier RJ. Cervical ripening with transcervical foley catheter and the risk of uterine rupture. Obstet Gynecol. 2004 Jan;103(1):18-23. doi: 10.1097/01.AOG.0000109148.23082.C1. PMID 14704239
- [Background] Carbone JF, Tuuli MG, Fogertey PJ, Roehl KA, Macones GA. Combination of Foley bulb and vaginal misoprostol compared with vaginal misoprostol alone for cervical ripening and labor induction: a randomized controlled trial. Obstet Gynecol. 2013 Feb;121(2 Pt 1):247-252. doi: 10.1097/AOG.0b013e31827e5dca. PMID 23303106
- [Background] Cromi A, Ghezzi F, Agosti M, Serati M, Uccella S, Arlant V, Bolis P. Is transcervical Foley catheter actually slower than prostaglandins in ripening the cervix? A randomized study. Am J Obstet Gynecol. 2011 Apr;204(4):338.e1-7. doi: 10.1016/j.ajog.2010.11.029. Epub 2011 Jan 26. PMID 21272849
- [Background] Delaney S, Shaffer BL, Cheng YW, Vargas J, Sparks TN, Paul K, Caughey AB. Labor induction with a Foley balloon inflated to 30 mL compared with 60 mL: a randomized controlled trial. Obstet Gynecol. 2010 Jun;115(6):1239-1245. doi: 10.1097/AOG.0b013e3181dec6d0. PMID 20502296
- [Background] Fitzpatrick CB, Grotegut CA, Bishop TS, Canzoneri BJ, Heine RP, Swamy GK. Cervical ripening with foley balloon plus fixed versus incremental low-dose oxytocin: a randomized controlled trial. J Matern Fetal Neonatal Med. 2012 Jul;25(7):1006-10. doi: 10.3109/14767058.2011.607522. Epub 2011 Dec 14. PMID 21793769
- [Background] Kashanian M, Nazemi M, Malakzadegan A. Comparison of 30-mL and 80-mL Foley catheter balloons and oxytocin for preinduction cervical ripening. Int J Gynaecol Obstet. 2009 May;105(2):174-5. doi: 10.1016/j.ijgo.2009.01.005. Epub 2009 Feb 20. No abstract available. PMID 19232606
- [Background] Levy R, Kanengiser B, Furman B, Ben Arie A, Brown D, Hagay ZJ. A randomized trial comparing a 30-mL and an 80-mL Foley catheter balloon for preinduction cervical ripening. Am J Obstet Gynecol. 2004 Nov;191(5):1632-6. doi: 10.1016/j.ajog.2004.03.033. PMID 15547534
- [Background] Moraes Filho OB, Albuquerque RM, Cecatti JG. A randomized controlled trial comparing vaginal misoprostol versus Foley catheter plus oxytocin for labor induction. Acta Obstet Gynecol Scand. 2010 Aug;89(8):1045-52. doi: 10.3109/00016349.2010.499447. PMID 20636243
- [Background] Pettker CM, Pocock SB, Smok DP, Lee SM, Devine PC. Transcervical Foley catheter with and without oxytocin for cervical ripening: a randomized controlled trial. Obstet Gynecol. 2008 Jun;111(6):1320-6. doi: 10.1097/AOG.0b013e31817615a0. PMID 18515515
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264
- [Derived] Gagnon J, Corlin T, Berghella V, Hoffman MK, Sciscione A, Marie PS, Schoen CN. Intracervical Foley catheter with and without oxytocin for labor induction with Bishop score </=3: a secondary analysis. Am J Obstet Gynecol MFM. 2021 Jul;3(4):100350. doi: 10.1016/j.ajogmf.2021.100350. Epub 2021 Mar 20. PMID 33757937
- [Derived] Schoen CN, Grant G, Berghella V, Hoffman MK, Sciscione A. Intracervical Foley Catheter With and Without Oxytocin for Labor Induction: A Randomized Controlled Trial. Obstet Gynecol. 2017 Jun;129(6):1046-1053. doi: 10.1097/AOG.0000000000002032. PMID 28486381

RESULTS

PARTICIPANT FLOW:
Groups:
- Nulliparous - Foley Only: Nulliparous women randomized to receive Foley only treatment will have a 20 French latex or silicone Foley catheter placed by the provider in the method they are most comfortable (direct visualization or indirectly). Balloons will have the ability to accommodate up to 80 ml of fluid to avoid rupture. The Foley balloon with be instilled with 60 ml of saline. The end of the catheter is then taped to the medial aspect of the patient's thigh on tension. No additional ripening agents or oxytocin will be administered while the Foley is in place. If spontaneous expulsion has not occurred, the Foley will be removed after 12 hours. Oxytocin will be administered per Christiana Care protocol after Foley removal.
  Transcervical Foley catheter
- Nulliparous - Foley and Oxytocin: Nulliparous women randomized to receive Foley and oxytocin treatment will have a 20 French latex or silicone Foley catheter placed by the provider in the method they are most comfortable (direct visualization or indirectly). Balloons will have the ability to accommodate up to 80 ml of fluid to avoid rupture. The Foley balloon with be instilled with 60 ml of saline. The end of the catheter is then taped to the medial aspect of the patient's thigh on tension. If spontaneous expulsion has not occurred, the Foley will be removed after 12 hours. Oxytocin will be administered per Christiana Care protocol immediately after Foley placement.
  Oxytocin
  Transcervical Foley catheter
- Multi(Primi)Parous - Foley Only: Multiparous and primiparous women randomized to receive Foley only treatment will have a 20 French latex or silicone Foley catheter placed by the provider in the method they are most comfortable (direct visualization or indirectly). Balloons will have the ability to accommodate up to 80 ml of fluid to avoid rupture. The Foley balloon with be instilled with 60 ml of saline. The end of the catheter is then taped to the medial aspect of the patient's thigh on tension. No additional ripening agents or oxytocin will be administered while the Foley is in place. If spontaneous expulsion has not occurred, the Foley will be removed after 12 hours. Oxytocin will be administered per Christiana Care protocol after Foley removal.
  Transcervical Foley catheter
- Multi(Primi)Parous - Foley and Oxytocin: Multiparous and primiparous women randomized to receive Foley and oxytocin treatment will have a 20 French latex or silicone Foley catheter placed by the provider in the method they are most comfortable (direct visualization or indirectly). Balloons will have the ability to accommodate up to 80 ml of fluid to avoid rupture. The Foley balloon with be instilled with 60 ml of saline. The end of the catheter is then taped to the medial aspect of the patient's thigh on tension. If spontaneous expulsion has not occurred, the Foley will be removed after 12 hours. Oxytocin will be administered per Christiana Care protocol immediately after Foley placement.
  Oxytocin
  Transcervical Foley catheter
Period: Overall Study
Arm/Group | Nulliparous - Foley Only | Nulliparous - Foley and Oxytocin | Multi(Primi)Parous - Foley Only | Multi(Primi)Parous - Foley and Oxytocin
Started | 94 | 90 | 67 | 72
Completed | 94 | 90 | 67 | 71
Not Completed | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nulliparous - Foley Only | Nulliparous - Foley and Oxytocin | Multi(Primi)Parous - Foley Only | Multi(Primi)Parous - Foley and Oxytocin | Total
Number analyzed (Participants) | 94 | 90 | 67 | 71 | 322
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (5) | 27 (6) | 31 (5) | 31 (5) | 29 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 90 | 67 | 71 | 322
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Asian | 6 | 3 | 3 | 0 | 12
  Race/Ethnicity: Black or African American | 41 | 30 | 39 | 35 | 145
  Race/Ethnicity: Caucasian | 38 | 49 | 16 | 29 | 132
  Race/Ethnicity: Hispanic | 7 | 5 | 8 | 5 | 25
  Race/Ethnicity: Other | 2 | 3 | 1 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Delivery Rate
Description: The rate of women who deliver in less than or equal to 24 hours from Foley placement.
Time Frame: Within 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Nulliparous - Foley Only | Nulliparous - Foley and Oxytocin | Multi(Primi)Parous - Foley Only | Multi(Primi)Parous - Foley and Oxytocin
Number analyzed (Participants) | 94 | 90 | 67 | 71
Participants | 40 | 58 | 48 | 62

2. Secondary Outcome: Number of Participants With Time to Delivery Achieved Within 12 Hours
Description: Number of participants with a time from Foley placement to delivery less than or equal to 12 hours
Time Frame: Within 12 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Nulliparous - Foley Only | Nulliparous - Foley and Oxytocin | Multi(Primi)Parous - Foley Only | Multi(Primi)Parous - Foley and Oxytocin
Number analyzed (Participants) | 94 | 90 | 67 | 71
Participants | 2 | 7 | 13 | 23

3. Secondary Outcome: Total Time to Delivery
Time Frame: On average, 24-36 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nulliparous - Foley Only | Nulliparous - Foley and Oxytocin | Multi(Primi)Parous - Foley Only | Multi(Primi)Parous - Foley and Oxytocin
Number analyzed (Participants) | 94 | 90 | 67 | 71
hours | 26.1 [20.5 to 33.7] | 20.9 [16.2 to 27] | 18.6 [13.5 to 25.2] | 14.9 [10.7 to 21]

4. Secondary Outcome: Time to Foley Expulsion
Time Frame: 0-12 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nulliparous - Foley Only | Nulliparous - Foley and Oxytocin | Multi(Primi)Parous - Foley Only | Multi(Primi)Parous - Foley and Oxytocin
Number analyzed (Participants) | 94 | 90 | 67 | 71
hours | 11.8 [7.8 to 12.3] | 7.2 [4.8 to 11.8] | 7.9 [4.5 to 12] | 5.8 [4.1 to 8.4]

5. Secondary Outcome: Number of Vaginal Deliveries
Time Frame: Assessed after delivery, on average occurring between 24-48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Nulliparous - Foley Only | Nulliparous - Foley and Oxytocin | Multi(Primi)Parous - Foley Only | Multi(Primi)Parous - Foley and Oxytocin
Number analyzed (Participants) | 94 | 90 | 67 | 71
Participants | 59 | 49 | 54 | 59

6. Secondary Outcome: Regional Analgesia
Description: Regional analgesia used during Foley ripening
Time Frame: Assessed during the induction, labor and delivery period, on average occurring between 24-48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Nulliparous - Foley Only | Nulliparous - Foley and Oxytocin | Multi(Primi)Parous - Foley Only | Multi(Primi)Parous - Foley and Oxytocin
Number analyzed (Participants) | 94 | 90 | 67 | 71
Participants | 2 | 13 | 1 | 11

7. Secondary Outcome: Obstetric Complications
Time Frame: Assessed during induction, labor, delivery, and postpartum. On average, this would be over a 3-7 day time period
Measure: Count of Participants; unit: Participants
Arm/Group | Nulliparous - Foley Only | Nulliparous - Foley and Oxytocin | Multi(Primi)Parous - Foley Only | Multi(Primi)Parous - Foley and Oxytocin
Number analyzed (Participants) | 94 | 90 | 67 | 71
Participants
  Tachysystole | 8 | 10 | 1 | 3
  Chorioamnionitis | 17 | 11 | 3 | 2
  Meconium | 14 | 20 | 8 | 5
  Postpartum hemorrhage | 14 | 11 | 8 | 6
  Uterine rupture | 0 | 0 | 0 | 0
  Maternal death | 0 | 0 | 0 | 0

8. Secondary Outcome: Neonatal Outcome: NICU (Neonatal Intensive Care Unit) Admission, 5 Minutes Apgar <7
Time Frame: Assessed from birth through discharge, on average 2 days after birth
Measure: Count of Participants; unit: Participants
Arm/Group | Nulliparous - Foley Only | Nulliparous - Foley and Oxytocin | Multi(Primi)Parous - Foley Only | Multi(Primi)Parous - Foley and Oxytocin
Number analyzed (Participants) | 94 | 90 | 67 | 71
Participants
  NICU admission | 27 | 23 | 12 | 11
  5-minute Apgar score <7 | 5 | 0 | 2 | 1
  Macrosomia | 9 | 8 | 3 | 6

9. Secondary Outcome: Neonatal Outcome: Neonatal Weight
Time Frame: Assessed from birth through discharge, on average 2 days after birth
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Nulliparous - Foley Only | Nulliparous - Foley and Oxytocin | Multi(Primi)Parous - Foley Only | Multi(Primi)Parous - Foley and Oxytocin
Number analyzed (Participants) | 94 | 90 | 67 | 71
grams | 3301 (524) | 3278 (570) | 3177 (523) | 3164 (579)

ADVERSE EVENTS:
Arm/Group | Nulliparous - Foley Only | Nulliparous - Foley and Oxytocin | Multi(Primi)Parous - Foley Only | Multi(Primi)Parous - Foley and Oxytocin
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/90 | 0/67 | 0/71
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/90 | 0/67 | 0/71
Other Adverse Events (participants affected / at risk) | 1/94 | 0/90 | 0/67 | 1/71
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nulliparous - Foley Only (N=94) | Nulliparous - Foley and Oxytocin (N=90) | Multi(Primi)Parous - Foley Only (N=67) | Multi(Primi)Parous - Foley and Oxytocin (N=71)
Foley balloon rupture (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes